CLINICAL TRIAL: NCT01525849
Title: Randomized Evaluation of Maxillary Antrostomy Versus Ostial Dilation Efficacy Through Long-Term Follow-Up
Acronym: REMODEL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Entellus Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1984-001
Record Dates: First submitted 2012-02-01; First posted 2012-02-03 (Estimated); Results first posted 2017-02-24 (Actual); Last update posted 2017-02-24 (Actual); Status verified 2017-01

CONDITIONS: Chronic Sinusitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Balloon Sinus Dilation (Active Comparator): XprESS Multi-Sinus Dilation Balloon, FinESS Sinus Treatment
  Interventions: Device: Balloon Sinus Dilation
- Functional Endoscopic Sinus Surgery (Active Comparator): Traditional endoscopic sinus surgery (maxillary antrostomy and uncinectomy with optional anterior ethmoidectomy) using cutting, grasping, and microdebrider tools.
  Interventions: Procedure: Functional Endoscopic Sinus Surgery

INTERVENTIONS:
Device: Balloon Sinus Dilation — Balloon sinus dilation using the XprESS Multi-Sinus Dilation Tool or the FinESS SInus Treatment
  Arms: Balloon Sinus Dilation
Procedure: Functional Endoscopic Sinus Surgery — Endoscopic sinus surgery, specifically, maxillary antrostomy and uncinectomy with optional anterior ethmoidectomy
  Arms: Functional Endoscopic Sinus Surgery

SUMMARY:
The objective of this study is to show that long-term symptom improvement after sinus balloon dilation is not worse than symptom improvement after functional endoscopic sinus surgery (FESS) and that fewer postoperative debridements are required after balloon dilation than after FESS.

DETAILED DESCRIPTION:
This is a postmarket, multicenter, prospective, randomized clinical trial conducted at up to 15 US clinical sites comparing the efficacy of balloon sinus dilation with traditional endoscopic sinus surgery. The primary hypotheses were to demonstrate that: 1) long-term change in sinus symptoms after balloon dilation is not worse (non-inferior) than after FESS, and 2) balloon dilation is superior to FESS for a reduction in the number of postoperative debridements per patient. A minimum of 36 participants per arm is required to test the primary hypotheses. All participants will be followed through a minimum of 12 months post treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* maxillary sinus disease
* chronic sinusitis

Exclusion Criteria:

* fungal disease
* Samter's triad
* hemophilia
* prior sinus surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2011-12; Primary Completion 2014-02 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Entellus Medical, Plymouth, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Cutler J, Bikhazi N, Light J, Truitt T, Schwartz M; REMODEL Study Investigators. Standalone balloon dilation versus sinus surgery for chronic rhinosinusitis: a prospective, multicenter, randomized, controlled trial. Am J Rhinol Allergy. 2013 Sep-Oct;27(5):416-22. doi: 10.2500/ajra.2013.27.3970. Epub 2013 Aug 5. PMID 23920419
- [Result] Bikhazi N, Light J, Truitt T, Schwartz M, Cutler J; REMODEL Study Investigators. Standalone balloon dilation versus sinus surgery for chronic rhinosinusitis: a prospective, multicenter, randomized, controlled trial with 1-year follow-up. Am J Rhinol Allergy. 2014 Jul-Aug;28(4):323-9. doi: 10.2500/ajra.2014.28.4064. Epub 2014 May 12. PMID 24823902
- [Result] Chandra RK, Kern RC, Cutler JL, Welch KC, Russell PT. REMODEL larger cohort with long-term outcomes and meta-analysis of standalone balloon dilation studies. Laryngoscope. 2016 Jan;126(1):44-50. doi: 10.1002/lary.25507. Epub 2015 Jul 30. PMID 26228589

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened, randomized, treated, and followed at 14 US centers from June 2011 to May 2014.
Pre-assignment Details: After screening, informed consent, and baseline measures, participants were randomized 1:1 to balloon sinus dilation or FESS. The assigned procedure was to be performed within 60 days of randomization.
Groups:
- Balloon Sinus Dilation: Balloon sinus dilation using XprESS Multi-Sinus Dilation Balloon or FinESS Sinus Treatment
Period: Overall Study
Arm/Group | Balloon Sinus Dilation | Functional Endoscopic Sinus Surgery
Started | 76 | 75
Treated | 74 (2 withdrew before treatment: 1 didn't want balloon dilation, 1 unrelated medical issue.) | 61 (14 withdrew before treatment: 8 didn't want FESS, 1 too busy, 2 medical issues, 3 excl. criteria.)
6-Months | 73 | 60
Completed | 71 | 59
Not Completed | 5 | 16
Not completed — Lost to Follow-up | 3 | 2
Not completed — Withdrawal by Subject | 1 | 9
Not completed — Unrelated medical issue (not treated) | 1 | 2
Not completed — Anatomic exclusion criteria identified | 0 | 3

BASELINE CHARACTERISTICS:
Population: All treated participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Balloon Sinus Dilation | Functional Endoscopic Sinus Surgery | Total
Number analyzed (Participants) | 74 | 61 | 135
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (13.6) | 47.8 (14.1) | 46.9 (13.8)
Gender [Count of Participants; unit: Participants]
  Female | 48 | 36 | 84
  Male | 26 | 25 | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 5 | 11
  Not Hispanic or Latino | 68 | 56 | 124
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 1 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 65 | 56 | 121
  More than one race | 3 | 0 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 74 | 61 | 135
Sino-Nasal Outcome Test (SNOT-20) overall score [Mean (Standard Deviation); unit: units on a scale] — A validated patient-reported survey of 20 items related to sinonasal symptoms and severity assessed over the previous 2 weeks. Each item is scored from 0 (no problem) to 5 (problem as bad as it can be). The individual item scores are averaged to provide an overall score that ranges from 0 (best) to 5 (worst).
  units on a scale | 2.49 (0.88) | 2.52 (0.83) | 2.50 (0.85)

OUTCOME MEASURES:

1. Primary Outcome: Sinus Symptom Improvement
Description: Change from baseline in overall 20-item Sino-Nasal Outcome Test (SNOT-20) score. The SNOT-20 is a validated patient reported survey of 20 items related to sinonasal symptoms and severity assessed over the previous 2 weeks. Each item is scored from 0 (no problem) to 5 (problem as bad as it can be). The individual item scores are averaged to provide and overall score that ranges from 0 (best) to 5 (worst).
Time Frame: Baseline and 1-year
Population: All treated participants with matched pair SNOT-20 data at baseline and 1-year.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Balloon Sinus Dilation | Functional Endoscopic Sinus Surgery
Number analyzed (Participants) | 69 | 58
units on a scale
  Change from baseline | -1.59 (1.08) | -1.60 (1.00)
  Mean overall SNOT-20 score at 1-year | 0.88 (0.91) | 0.88 (0.76)
Statistical Analysis 1: Comparison: Balloon Sinus Dilation vs Functional Endoscopic Sinus Surgery; Non-inferiority test to demonstrate that the long-term (1-year) change in sinus symptoms (overall SNOT-20 score) after balloon dilation is not worse than after FESS; Test type: Non-Inferiority or Equivalence — Significance level=0.025 (1-sided alpha), power=90%, delta=0.8, true difference=0, SD for both arms=1.0. A total sample size of 72 participants (36 per arm) was required to test the hypothesis; p < 0.001, t-test, 1 sided

2. Primary Outcome: Debridements
Description: Number of postoperative debridements per participant
Time Frame: 1-year
Population: All treated participants
Measure: Mean (Standard Deviation); unit: debridements per participant
Arm/Group | Balloon Sinus Dilation | Functional Endoscopic Sinus Surgery
Number analyzed (Participants) | 74 | 61
debridements per participant | 0.23 (0.65) | 1.03 (0.87)
Statistical Analysis 1: Comparison: Balloon Sinus Dilation vs Functional Endoscopic Sinus Surgery; Test for superiority of balloon dilation over FESS. Significance level=0.025 (1-sided alpha), power=90%, BD estimate=0.5, FESS estimate=1.5, SD for both arms=1.0. A total sample size of 46 participants (23 per arm) was required to test the hypothesis; Test type: Superiority or Other; p < 0.0001, t-test, 1 sided

3. Secondary Outcome: Revision Rate
Description: Number of participants requiring repeat sinus procedures
Time Frame: 1-year
Population: All treated participants with 1-year follow-up (or a revision surgery before 1-year follow-up if no 1-year follow-up).
Measure: Count of Participants; unit: Participants
Arm/Group | Balloon Sinus Dilation | Functional Endoscopic Sinus Surgery
Number analyzed (Participants) | 71 | 59
Participants | 1 | 1
Statistical Analysis 1: Comparison: Balloon Sinus Dilation vs Functional Endoscopic Sinus Surgery; Test type: Superiority or Other; p = 0.628, t-test, 2 sided

4. Secondary Outcome: Complication Rate
Description: Number of participants experiencing 1 or more serious adverse events related to the device and/or procedure
Time Frame: Duration of study (minimum of 12 months)
Population: All randomized participants
Measure: Count of Participants; unit: Participants
Arm/Group | Balloon Sinus Dilation | Functional Endoscopic Sinus Surgery
Number analyzed (Participants) | 76 | 75
Participants | 0 | 0

5. Secondary Outcome: Recovery Time
Description: Mean time (days) after procedure for participants to return to normal activities
Time Frame: 6-months
Population: All treated participants with 6-month follow-up.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Balloon Sinus Dilation | Functional Endoscopic Sinus Surgery
Number analyzed (Participants) | 73 | 60
days | 1.7 (1.3) | 5.0 (5.9)
Statistical Analysis 1: Comparison: Balloon Sinus Dilation vs Functional Endoscopic Sinus Surgery; Test type: Superiority or Other; p < 0.0001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Duration of study (minimum of 1-year) for all treated participants.
Description: Participants continued to be followed every 6 months after completion of the 1-year follow-up until all participants had completed the 1-year follow-up. Adverse events were collected at all follow-up visits. Adverse events occurring after randomization for participants who did not undergo treatment are included until the time of their withdrawal.
Arm/Group | Balloon Sinus Dilation | Functional Endoscopic Sinus Surgery
Serious Adverse Events (participants affected / at risk) | 1/76 | 2/75
Other Adverse Events (participants affected / at risk) | 0/76 | 0/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Balloon Sinus Dilation (N=76) | Functional Endoscopic Sinus Surgery (N=75)
Acute Gastroenteritis (Gastrointestinal disorders) | 1 (1) | 0 (0) — Gastoenteritis reported at 118 days post procedure (unrelated).
Atypical Chest Pain (Cardiac disorders) | 0 (0) | 1 (1) — Participant underwent tests to rule out coronary artery disease. Participant withdrew before study procedure (unrelated).
Infection (Infections and infestations) | 0 (0) | 1 (1) — Methicillin-resistant Staph aureus infection and cellulitis on the nasal tip reported at 276 days post procedure (unrelated).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less